CLINICAL TRIAL: NCT03623763
Title: Vitamin D Level Among Water Sports Elite Athletes in Uzbekistan
Brief Title: Vitamin D Level Among Athletes in Uzbekistan
Status: Suspended | Type: Observational
Why Stopped: Financial difficulities
Sponsor: Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan (Other Government)
Responsible Party: Principal Investigator, Svetlana Osipova, MD, PhD, DS, Senior researcher, Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan
Other Study IDs: #30072018
Record Dates: First submitted 2018-07-29; First posted 2018-08-09 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Athletes; Respiratory Infection; Cytokines; Vitamin D
Keywords: vitamin D; water sport; IL-4; IL-6; TNF-a; IFN-gamma; athletes; respiratory infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy individuals: Individuals without any complaints and chronic diseases
  Interventions: Diagnostic Test: Serologic tests of blood samples
- Swimmers: Elite athletes - swimmers to distance of national team of Uzbekistan
  Interventions: Diagnostic Test: Serologic tests of blood samples
- Synchronized swimmers: Elite athletes - swimmers of national team of Uzbekistan
  Interventions: Diagnostic Test: Serologic tests of blood samples

INTERVENTIONS:
Diagnostic Test: Serologic tests of blood samples — Five milliliters of peripheral venous blood will be (after 8-12 hours of fasting) from each participant and will be collected into Human Tube Serum Gel - C/A for ELISA. All blood samples will be collected in August and January. Serum levels of 25(OH) VD and TNF-α, IFN-γ, IL-4 and IL-6 will be detected by ELISA technique

SUMMARY:
The purpose of the study is to determine vitamin D (VD) levels and upper respiratory tract infections (URTI) morbidity among elite athletes engaged in water sports in Uzbekistan. Serum levels of 25(OH) VD and TNF-α, IFN-γ, IL-4 and IL-6 will be detected by ELISA technique among elite athletes and control population in spring and autumn.

DETAILED DESCRIPTION:
Study center The prospective diagnostic study will be conducted on the basis of Uzbek State University of Physical Education and Sport and Research Institute of Epidemiology, Microbiology and Infectious Diseases, Tashkent, Uzbekistan during the period from January 2017 till January 2019.

Both informed and written consents will be obtained from the athletes and healthy individuals.

Study participants Aproximately 40 elite athletes engaged in water sport and 60 healthy individuals will be included to the study.

All the participants will be residents of Uzbekistan.

Serological tests Five milliliters of peripheral venous blood will be taken (after 8-12 hours of fasting) from each participant and will be collected into Human Tube Serum Gel - C/A for ELISA. All blood samples will be collected in August and January.

Serum levels of 25(OH) VD and TNF-α, IFN-γ, IL-4 and IL-6 will be detected by ELISA technique.

Enzyme immunoassay for the quantitative measurement of total 25-OH-Vitamin D (Vitamin D2 and D3) in human serum.

Solid phase enzyme-linked immunosorbent assay (ELISA) based on the competition principle. An unknown amount of antigen present in the sample and a fixed amount of enzyme labelled antigen compete for the binding sites of the antibodies coated onto the wells. After incubation the wells are washed to stop the competition reaction. After the substrate reaction the intensity of the developed colour is inversely proportional to the amount of the antigen in the sample. Results of samples can be determined directly using the standard curve.

A sandwich enzyme immunoassay for in vitro quantitative measurement of TNFa The microplate provided in this kit has been pre-coated with an antibody specific to TNFa. Standards or samples are then added to the appropriate microplate wells with a biotin-conjugated antibody specific to TNFa. Next, Avidin conjugated to Horseradish Peroxidase (HRP) is added to each microplate well and incubated. After TMB substrate solution is added, only those wells that contain TNFa, biotin-conjugated antibody and enzyme-conjugated Avidin will exhibit a change in color. The enzyme-substrate reaction is terminated by the addition of sulphuric acid solution and the color change is measured spectrophotometrically at a wavelength of 450nm ± 10nm. The concentration of TNFa in the samples is then determined by comparing the O.D. of the samples to the standard curve.

IFN-γ, IL-4 and IL-6 will be detected and measured by the same enzyme immunoassay method presented above.

Data analysis will be performed with the program Origin 6.1 (OriginLab, Northampton, MA).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Swimmers to distance
* Synchronized swimmers

Exclusion Criteria:

* chronic infectious and noninfectious diseases
* acute infectious and noninfectious diseases
* history of using VD supplements within six months or drugs usage within three months.

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy individuals Swimmers to distance Synchronized swimmers
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Vitamin D level in elite athletes | up to 36 months
  In this study we expect to determine of serum level of vitamin D in elite athletes of Uzbekistan
Correlation between cytokine status (TNF-α, IFN-γ, IL-4 and IL-6 ) and vitamin D level among elite athletes | up to 36 months
  In this study we expect to find association between cytokine status and vitamin D level in elite athletes.
Incidence of upper respiratory infection among elite athletes with vitamin D deficiency/insufficiency/sufficiency | up to 36 months
  In this study we expect to find a role of vitamin D in development of upper respiratory infection among elite athletes.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Umarov J, Kerimov F, Toychiev A, Davis N, Osipova S. Association of the 25(OH) vitamin D status with upper respiratory tract infections morbidity in water sports elite athletes. J Sports Med Phys Fitness. 2019 Dec;59(12):2058-2065. doi: 10.23736/S0022-4707.19.09834-7. Epub 2019 May 2. PMID 31062952
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31062952/